CLINICAL TRIAL: NCT01900496
Title: Pilot Study of Rituximab and Brentuximab Vedotin With Deferred BMT for Relapsed Classical Hodgkin Lymphoma
Brief Title: Study of Rituximab and Brentuximab Vedotin for Relapsed Classical Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1354; NA_00080336 (Other: JHM IRB)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma
Keywords: cHL; Hodgkin lymphoma; Lymphoma; relapsed Lymphoma; SGN-35; Brentuximab Vedotin; Rituxan; Rituximab
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Brentuximab Vedotin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab vedotin & Rituximab (Experimental): Brentuximab vedotin:
  Will be administered at 1.8 mg/kg IV over 30 minutes is given for up to 10 doses (cycles), with a cycle length of 21 days. Brentuximab vedotin is first given on day 1 of cycles 1, 2, 3, and 4 as a single agent (weeks 0, 3, 6, and 9, respectively). Four cycles are chosen because of the 12-week median time to CR in the pivotal phase 2 trial of brentuximab vedotin after autologous BMT for HL.
  Brentuximab vedotin will be administered with Rituximab at 375 mg/m2 IV is given for up to 8 "induction" doses: day 1 of week 6, 7, 8, and 9; day 1 of week 12, 15, 18 and 21. This is followed by rituximab "maintenance" (375 mg/m2 IV once every 3 months x 2 doses) to complete a ~ 1 year total course of therapy.
  Interventions: Biological: Brentuximab vedotin; Biological: Rituximab

INTERVENTIONS:
Biological: Brentuximab vedotin — Day 1 every three weeks (weeks 0, 3, 6, 9, ... 27): 1.8 mg/kg IV. Ten doses maximum.
  Other Names: SGN-35; Adcetris
Biological: Rituximab — Day 1 of weeks 12, 13, 14, 15, 18, 21, 24, and 27: 375 mg/m^2 IV. Additional doses are given at three and six months post week 27.
  Other Names: Rituxan

SUMMARY:
This research is being done to study a combination of Brentuximab vedotin and Rituximab for the treatment of relapsed Hodgkin's Lymphoma (HL).

DETAILED DESCRIPTION:
This research is being done to study a combination of drugs for relapsed Hodgkin's Lymphoma (HL) that may be easier to tolerate than standard therapies and that does not involve an autologous blood or marrow transplant (BMT, also called a stem cell transplant).The study is for people with HL who have never received treatment for relapsed lymphoma, except for radiation therapy. Usually, when HL relapses for the first time, the standard is to receive combinations of chemotherapy, including an autologous blood or marrow transplant (BMT, also called a stem cell transplant) which has about a 40% cure rate. BMT may cure the HL, but also may be associated with serious side effects and risks. This research looks at a combination of drugs for relapsed HL that may not have the side effects of standard therapies and that does not involve BMT. The goal is to treat the lymphoma effectively with drugs that we expect will have fewer side effects, while avoiding a treatment like BMT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Biopsy-proven diagnosis of classical Hodgkin Lymphoma (regardless of HRS cell CD20 expression) per the World Health Organization classification criteria24; lymphocyte predominant histology is excluded
* Untreated relapse of classical Hodgkin Lymphoma (with the exception of steroids) as follows:HL that relapsed > 3 months after completion of first-line chemotherapy or combined modality therapy, and has not yet been treated with salvage chemotherapy, Stage I-II HL that relapsed > 3 months after first-line chemotherapy, then relapsed after radiation therapy delivered with curative intent, and has not yet been treated with salvage chemotherapy
* Radiographically measurable disease (> 1 focus of lymphoma measuring > 1.5 cm)
* Baseline laboratories: ANC > 1000/uL and platelets > 75,000/uL, unless due to bone marrow involvement by lymphoma, Serum creatinine < 2.0 mg/dL, Total bilirubin < 2.0 mg/dL (excluding Gilbert's syndrome), unless due to lymphoma
* ECOG performance status 0, 1 or 2.

Exclusion Criteria:

* Active concurrent malignancy with the exception of superficial non-melanoma skin cancer and cervical carcinoma in situ.
* Primary induction failure, defined as failure to achieve CR with first-line chemotherapy or chemoradiation, disease progression during first-line chemotherapy or chemoradiation, or progression or biopsy-proven disease persistence within 8 weeks of first-line therapy completion
* Prior brentuximab vedotin or rituximab for lymphoma
* Grade > 2 peripheral neuropathy
* HIV infection, active hepatitis B infection, or active hepatitis C infection

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Failure-free survival | Up to 7 months
  Percentage of participants alive without any of the following: death, disease progression or relapse, or failure to achieve complete remission as defined by the Cheson criteria. Per Cheson Criteria: Complete Response (CR) is disappearance of all evidence of disease; Partial Response (PR) is regression of measurable disease and no new sites (≥50% decrease in sum of product diameters of up to 6 largest dominant masses and splenic/liver nodules), and no increase in size of other nodes/liver/spleen; reduction in target lesions, no growth of non-target or new lesions; Progression is any new lesion or increase by ≥50% of previously involved sites from the nadir

SECONDARY OUTCOMES:
Safety of combination of brentuximab vedotin and rituximab in relapsed classical Hodgkin's Lymphoma | Up to 7 months
  Percentage of participants with grade 3-4 adverse events by CTCAE 4.0.
Survival | Up to 7 months
  Percentage of participants alive with and without disease relapse.
Response rate | Up to 7 months
  Percentage of participants with partial and complete remissions as defined by Cheson criteria: Complete Response (CR) is disappearance of all evidence of disease; Partial Response (PR) is regression of measurable disease and no new sites (≥50% decrease in sum of product diameters of up to 6 largest dominant masses and splenic/liver nodules), and no increase in size of other nodes/liver/spleen; reduction in target lesions, no growth of non-target or new lesions
Time to best response | Up to 7 months
  Median number of weeks from protocol initiation to best response.
Duration of response | Up to 7 months
  Median number of weeks that best response was maintained until disease relapse or death.
Measurement of circulating clonotypic B cells (CCBCs) | Pre-study, Day 1, Week 12, Week 18, Week 24, Week 30, and time of relapse
  Median percentage change in CCBCs between initiation and completion of study.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Wagner-Johnston, MD, Principal Investigator — The Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Canceer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT01900496/Prot_SAP_000.pdf